CLINICAL TRIAL: NCT06725030
Title: PRECISE: A Post-market, Real-world Experience: Expanding Access to Care by Incorporating the Symani® Surgical System and Enabling Surgeons
Brief Title: A Post-market, Real-world Experience: Expanding Access to Care by Incorporating the Symani® Surgical System and Enabling Surgeons
Acronym: PRECISE
Status: Recruiting | Type: Observational
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Other Study IDs: CDC-00136
Record Dates: First submitted 2024-12-05; First posted 2024-12-09 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Open Surgery; Lymphedema; Free Tissue Transfer; Microsurgery; Anastomosis, Surgical
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Free Tissue Transfer Surgery
  Interventions: Device: Symani Surgical System
- Lymphovenous Anastomosis Surgery
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — The Symani Surgical System (Symani) is designed for open microsurgery procedures, featuring articulated and interchangeable instruments.

SUMMARY:
The objective of this study is to evaluate the Symani System's safety and effectiveness for microsurgical anastomosis during free tissue transfer surgery and lymphovenous anastomosis surgery.

The primary endpoints are:

* Effectiveness- Rate of intraoperative anastomosis patency at first attempt.
* Safety- Freedom from device-related adverse events.

Participants will receive treatment as standard of care and be asked to:

* Allow the researchers to access and use their information.
* If participants are undergoing a lymphedema procedure, they will be asked to undergo a questionnaire as part of the study.
* Participants will be asked to comply with the follow-up visits and complete all study procedures/questionnaires as outlined in the protocol.

ELIGIBILITY:
Pre Operative Inclusion Criteria:

1. At least 22 years of age
2. Patient agrees to participate in the study, return for all required follow-up visits, complete all study procedures, and has willingly provided written informed consent after receiving all information related to the study, its requirements, and the robotic assisted procedure
3. Patient has a clinical indication for a microsurgical anastomosis of vessels between 0.1 and 2.5 mm in conjunction with open free-flap surgery of the breast or extremities and/or lymphovenous anastomosis surgery of the extremities
4. Investigator deems the candidate acceptable for free flap transfer surgery and/or lymphovenous anastomosis surgery with a robotic assisted microsurgical anastomosis in accordance with the Symani System's Instructions for Use (IFU)

Cohort Specific Pre- Operative Inclusion Criteria:

Free Tissue Transfer Surgery: N/A

Lymphovenous Anastomosis Surgery

1. Swelling of one limb that is not completely reversed by elevation or compression
2. Stage I-II lymphedema at screening, based on the International Society of Lymphology (ISL) staging system
3. At least one of the following positive quantitative measurements:

   1. Volumetry differential between affected limb and contralateral limb must be at least 10% of the other
   2. Bioimpedance (L-Dex) differential, if feasible, between affected limb and contralateral limb of at least 10 units
4. Completion of a full course of complete decongestive therapy (CDT), according to ISL guidelines, for at least 12 weeks prior to screening, including use of compression garments for at least 12 weeks without change in regimen
5. Willingness to comply with recommended regimen of self-care, with consistent use of appropriately sized compression garments from screening through the entire study duration (through the 3-month follow-up visit).

Pre-Operative Exclusion Criteria:

1. Patients who are incapable and/or unwilling to provide informed consent
2. Active systemic infection under treatment with intravenous antibiotics
3. Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders, previous mental disorders, or other disorders that may significantly affect the data collection or the ability to comply with the protocol per the investigators discretion
4. Known history of significant bleeding, coagulopathy, or Von Willebrand's disease
5. Patients with implanted pacemaker
6. Planned vein graft
7. Currently receiving chemotherapy or radiation therapy
8. History of chronic kidney disease
9. History of chronic liver disease
10. Currently enrolled in any other investigational clinical studies that the investigator believes may impact patient safety or outcomes
11. Patients belonging to vulnerable populations, such as pregnant women, or ineligible to participate for other reasons in the judgement of the investigator

Cohort Specific Pre-Operative Exclusion Criteria:

Free Tissue Transplant Surgery:

1. Patients with buried flaps
2. Multiple flaps planned for the procedure

Lymphovenous Anastomosis Surgery:

1. Patients > 75 years of age
2. Patients with prior lymphatic reconstruction surgery
3. Patients with venous edema (arising from increased capillary filtration)
4. Patients with other medical conditions that could lead to acute limb edema, such as (but not limited to) acute venous thrombosis or heart failure
5. Patients with other medical conditions that could result in symptoms which overlap symptoms of lymphedema
6. Current infection in the affected limb
7. Patients who experience more than one episode of cellulitis in a six month period over the past two years
8. Current evidence or a history of malignancy within the past 6 months (if the participant has undergone cancer treatment, this must have been completed > 6 months prior to enrollment)
9. Known iodine sensitivity
10. Patient's lymphatic disease is due to lipedema
11. Patients with bilateral lymphedema or lymphedema in multiple anatomical locations

Intra Operative Exclusion Criteria:

1. Any presenting condition discovered intraoperatively that, in the opinion of the investigator, would make participating in this study not in the patient's best interest
2. The patient does not have at least one robotic stitch attempted during the index procedure

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for the PRECISE Study will be adults with a clinical indication for a microsurgical anastomosis of vessels between 0.1 and 2.5 mm in conjunction with open free flap surgery of the breast or extremities and/or lymphovenous anastomosis surgery of the extremities.
Sampling Method: Probability Sample
Enrollment: 455 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Freedom from device-related adverse events from the start of the index procedure through 30-days post index procedure as adjudicated by a Clinical Events Committee | From participants index procedure through 30-days post index procedure.
  All adverse events will be evaluated from the start of the index procedure through 30-days post index procedure. Adverse events will be reviewed by a Clinical Events Committee (CEC) to determine probable or causal relationships with the device. All device-related serious adverse events will be summarized descriptively.
Intraoperative anastomosis patency at first attempt. | The duration of the participants index procedure.
  Intraoperative anastomosis patency will be measured for each robotic anastomosis per standard of care and will be evaluated after the first attempt of the anastomosis during the index procedure.

SECONDARY OUTCOMES:
Intraoperative anastomosis patency prior to closure. | The duration of participants index procedure.
  Intraoperative anastomosis patency prior to closure will be measured for each robotic anastomosis per standard of care and will be evaluated prior to closure of the procedure site during the index procedure.
Anastomosis suturing time (including robotic time and manual time). | The duration of participants index procedure.
  Anastomosis suturing time of the index procedure will be collected for each participant and summarized. Robotic anastomosis time and manual anastomosis time will be recorded for each anastomosis. For each anastomosis within an operation, the total suture time (robotic plus manual) will be derived as total robotic anastomosis time plus total manual anastomosis time.
Number of robotic and manual stitches per anastomosis. | The duration of participants index procedure.
  The number of robotic stitches placed and the number of manual stitches placed per anastomosis in the index procedure will be collected for each anastomosis and summarized. For each anastomosis within an operation, the total stitches placed (robotic plus manual) will be derived as total robotic stitches placed plus total manual stitches.
Procedure time. | The duration of participants index procedure.
  Procedure time of the index procedure will be collected for each participant and summarized. The incision start time and closure end time will be recorded. The procedural time will be derived from incision time subtracted from closure time.
Technical Success. | The duration of participants index procedure.
  Technical success is defined as freedom from device malfunction resulting in unplanned conventional suturing. Device malfunctions and the associated outcome will be collected. This endpoint will be evaluated throughout the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bohdan Pomahac, MD, Principal Investigator — Yale New Haven Medical Center
Locations (4):
- United States (4):
  - Cedars Sinai Medical Center, Beverly Hills, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic, Cleveland, Ohio